CLINICAL TRIAL: NCT03952585
Title: A Randomized Phase II/III Trial of De-Intensified Radiation Therapy for Patients With Early-Stage, P16-Positive, Non-Smoking Associated Oropharyngeal Cancer
Brief Title: De-intensified Radiation Therapy With Chemotherapy (Cisplatin) or Immunotherapy (Nivolumab) in Treating Patients With Early-Stage, HPV-Positive, Non-Smoking Associated Oropharyngeal Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-03015; NCI-2019-03015 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-HN005 (Other: NRG Oncology); NRG-HN005 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Results first posted 2025-05-02 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-06

CONDITIONS: Basaloid Squamous Cell Carcinoma; Clinical Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Clinical Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Oropharyngeal Squamous Cell Carcinoma; Papillary Squamous Cell Carcinoma; Pathologic Stage I HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Pathologic Stage II HPV-Mediated (p16-Positive) Oropharyngeal Carcinoma AJCC v8; Squamous Cell Carcinoma
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Squamous Cell | interventions — Biopsy; Specimen Handling; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Fluorodeoxyglucose F18; Radiotherapy, Image-Guided; Radiotherapy, Intensity-Modulated; Magnetic Resonance Spectroscopy; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (Standard RT + cisplatin) (Active Comparator): Patients undergo standard dose RT as 70 Gy IMRT or IGRT over 6 fractions per week and receive 100 mg/m^2/day cisplatin IV over 30-60 minutes on days 1 and 22. Treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients receive FDG and undergo PET/CT or CT during screening and during follow up, and undergo MRI during follow up. Patients may also undergo tissue biopsy and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Radiation: Image Guided Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (Reduced RT + cisplatin) (Experimental): Patients undergo reduced dose RT as 60 Gy IMRT or IGRT QD over 5 fractions per week and receive 100 mg/m^2/day cisplatin IV over 30-60 minutes on days 1 and 22. Treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients receive FDG and undergo PET/CT or CT during screening and during follow up, and undergo MRI during follow up. Patients may also undergo tissue biopsy and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Radiation: Image Guided Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Procedure: Magnetic Resonance Imaging; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm III (Reduced RT + nivolumab) (Experimental): Beginning 1 week prior to radiation, patients receive 240 mg fixed dose nivolumab IV over 30 minutes on day 1. Treatment repeats every 2 weeks (14 days) for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo reduced dose RT as 60 Gy IMRT or IGRT over 6 fractions per week for 5 weeks in the absence of disease progression or unacceptable toxicity. Patients receive FDG and undergo PET/CT or CT during screening and during follow up, and undergo MRI during follow up. Patients may also undergo tissue biopsy and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Other: Fludeoxyglucose F-18; Radiation: Image Guided Radiation Therapy; Radiation: Intensity-Modulated Radiation Therapy; Biological: Nivolumab; Procedure: Positron Emission Tomography; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tissue biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
  Arms: Arm I (Standard RT + cisplatin); Arm II (Reduced RT + cisplatin)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Other: Fludeoxyglucose F-18 — Receive FDG
  Other Names: 18FDG; FDG; Fludeoxyglucose (18F); fludeoxyglucose F 18; Fludeoxyglucose F18; Fluorine-18 2-Fluoro-2-deoxy-D-Glucose; Fluorodeoxyglucose F18
Radiation: Image Guided Radiation Therapy — Undergo IGRT
  Other Names: IGRT; Image Guided Radiotherapy; image-guided radiation therapy; Image-Guided Radiotherapy
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity modulated radiation therapy (procedure); Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
  Arms: Arm I (Standard RT + cisplatin); Arm II (Reduced RT + cisplatin)
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm III (Reduced RT + nivolumab)
Procedure: Positron Emission Tomography — Undergo PET
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II/III trial studies how well a reduced dose of radiation therapy works with nivolumab compared to cisplatin in treating patients with human papillomavirus (HPV)-positive oropharyngeal cancer that is early in its growth and may not have spread to other parts of the body (early-stage), and is not associated with smoking. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Chemotherapy drugs, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. This trial is being done to see if a reduced dose of radiation therapy and nivolumab works as well as standard dose radiation therapy and cisplatin in treating patients with oropharyngeal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To demonstrate non-inferiority in terms of progression-free survival (PFS) of concurrent reduced-dose radiation therapy (RT) with cisplatin or concurrent reduced-dose radiation therapy with nivolumab to the current standard of care (standard-dose RT with cisplatin). (Phase II) (Arm 2 [concurrent reduced-dose RT with cisplatin] was dropped after interim futility analysis in phase II.) II. To demonstrate non-inferiority in terms of progression-free survival (PFS) of concurrent reduced-dose radiation therapy (RT) with nivolumab to the current standard of care (standard-dose RT with cisplatin). (Phase II) III. To demonstrate co-primary endpoints of non-inferiority of PFS and superiority of quality of life (QOL) as measured by the MD Anderson Dysphagia Inventory (MDADI) of concurrent reduced-dose radiation with cisplatin or concurrent reduced-dose radiation with nivolumab to the current standard of care (standard-dose RT with cisplatin). (Phase III) (Arm 2 [concurrent reduced-dose RT with cisplatin] was dropped after interim futility analysis in phase II.) IV. To demonstrate co-primary endpoints of non-inferiority of PFS and superiority of quality of life (QOL) as measured by the MD Anderson Dysphagia Inventory [MDADI] of concurrent reduced-dose radiation with nivolumab to the current standard of care (standard-dose RT with cisplatin). (Phase III)

SECONDARY OBJECTIVES:

I. To compare patterns of failure (local and regional relapse versus distant) and overall survival between the experimental arm and the control arm.

II. To assess long term PFS, overall survival, and toxicity between the experimental arm and the control arm.

III. To determine acute and late toxicity profiles as measured by the Common Terminology Criteria for Adverse Events (CTCAE).

IV. To explore the symptomatic adverse events (AEs) for tolerability of each treatment arm as measured by the Patient-Reported Outcomes (PRO)-CTCAE.

V. To compare changes in patient-reported outcomes (Hearing Handicap Inventory for Adults-Screening [HHIA-S], European Organization for Research and Treatment of Cancer [EORTC]-Quality of Life Questionnaire [QLQ]30) between the experimental arm and the control arm.

VI. To assess the association of fludeoxyglucose F-18 (FDG)-positron emission tomography (PET)/computed tomography (CT) at baseline with locoregional control and PFS.

VII. To estimate the negative predictive value of the 12-14 weeks post-radiation therapy (RT) FDG-PET/CT in terms of locoregional control rates and PFS rates at 1 and 2 years.

EXPLORATORY OBJECTIVES:

I. To collect blood and tissue specimens for future translation research. II. To optimize radiotherapy treatment plan quality assurance methodology for radiotherapy planning and imaging.

III. To compare changes in patient-reported outcomes (European Quality of Life Five Dimension Five Level Scale [EQ-5D-5L]) between the experimental arm and the control arm.

IV. To collect Modified Barium Swallow (MBS) data for future review and analysis.

OUTLINE:

PHASE II: Patients are randomized to 1 of 3 arms.

ARM I: Patients undergo standard dose RT as 70 Gy intensity modulated radiation therapy (IMRT) or image-guided radiation therapy (IGRT) over 6 fractions per week and receive 100 mg/m^2/day cisplatin intravenously (IV) over 30-60 minutes on days 1 and 22. Treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients receive fludeoxyglucose F-18 (FDG) and undergo positron emission tomography (PET)/computed tomography (CT) or CT during screening and during follow up, and undergo magnetic resonance imaging (MRI) during follow up. Patients may also undergo tissue biopsy and blood sample collection throughout the study.

ARM II (CLOSED TO ACCRUAL 03-FEB-2023): Patients undergo reduced dose RT as 60 Gy IMRT or IGRT once daily (QD) over 5 fractions per week and receive 100 mg/m^2/day cisplatin IV over 30-60 minutes on days 1 and 22. Treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients receive FDG and undergo PET/CT or CT during screening and during follow up, and undergo MRI during follow up. Patients may also undergo tissue biopsy and blood sample collection throughout the study.

ARM III: Beginning 1 week prior to radiation, patients receive 240 mg fixed dose nivolumab IV over 30 minutes on day 1. Treatment repeats every 2 weeks (14 days) for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo reduced dose RT as 60 Gy IMRT or IGRT over 6 fractions per week for 5 weeks in the absence of disease progression or unacceptable toxicity. Patients receive FDG and undergo PET/CT or CT during screening and during follow up, and undergo MRI during follow up. Patients may also undergo tissue biopsy and blood sample collection throughout the study.

PHASE III: Patients are randomized to Arm I and/or Arm III.

After completion of study treatment, patients are followed up at 12-14 weeks, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) proven diagnosis of squamous cell carcinoma (including the histological variants papillary squamous cell carcinoma and basaloid squamous cell carcinoma but not neuroendocrine phenotype) of the oropharynx (tonsil, base of tongue, soft palate, or oropharyngeal walls); cytologic diagnosis from a cervical lymph node is sufficient in the presence of clinical evidence of a primary tumor in the oropharynx. Clinical evidence should be documented, may consist of palpation, imaging, or endoscopic evaluation, and should be sufficient to estimate the size of the primary (for T stage)
* Patients must have clinically or radiographically evident measurable disease at the primary site or at nodal stations. Simple tonsillectomy or local excision of the primary without removal of nodal disease is permitted, as is excision removing gross nodal disease but with intact primary site. Limited neck dissections retrieving =< 4 nodes are permitted and considered as non-therapeutic nodal excisions
* P16-positive based on local site immunohistochemical tissue staining (defined as greater than 70% strong diffuse nuclear or nuclear and cytoplasmic staining of tumor cells). Fine needle aspiration (FNA) biopsy specimens may be used as the sole diagnostic tissue. Centers are encouraged to contact the pathology chair for clarification

  * Note: Institutions must screen patients, whose tumors must be p16-positive by immunohistochemistry (IHC) in order to be eligible for the trial using a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory. A rigorous laboratory accreditation process similar to the United States (U.S.) CLIA certification, such as the provincial accreditation status offered by the Ontario Laboratory Accreditation (OLA) Program in Canada, the College of American Pathologists (CAP), or an equivalent accreditation in other countries, is acceptable. The p16-positive results must be reported on the pathology report being submitted
  * Note: If p16 result is equivocal, positive HPV deoxyribonucleic acid (DNA) test of tumor specimen is acceptable and fulfills the eligibility criteria
* Clinical stage T1-2, N1, M0 (American Joint Committee on Cancer [AJCC], 8th edition [ed.]) or T3, N0-N1, M0 (AJCC, 8th ed.) including no distant metastases based on the following diagnostic workup:

  * General history and physical examination within 56 days prior to registration;
  * Exam with laryngopharyngoscopy (mirror or in office direct procedure acceptable) within 70 days prior to registration;
  * One of the following imaging studies is required within 56 days prior to registration:

    * FDG-PET/CT of the neck and chest (with or without contrast); FDG-PET/CT scan is strongly preferred and highly recommended to be used for eligibility OR
    * Chest CT (with or without contrast)
  * One of the following imaging studies is required within 28 days prior to registration:

    * A diagnostic CT scan of neck (with contrast and of diagnostic quality) OR
    * An magnetic resonance imaging (MRI) of the neck (with contrast and of diagnostic quality)
    * Note: A diagnostic quality CT or MRI with contrast or FDG-PET/CT scan of neck performed for the purposes of radiation planning may serve as both staging and planning tools
* Patients must provide their personal smoking history prior to registration. The lifetime cumulative history cannot exceed 10 pack-years. The following formula is used to calculate the pack-years during the periods of smoking in the patient's life; the cumulative total of the number of pack-years during each period of active smoking is the lifetime cumulative history

  * Number of pack-years = [Frequency of smoking (number of cigarettes per day) x duration of cigarette smoking (years)] / 20
  * Note: Twenty cigarettes is considered equivalent to one pack. The effect of non-cigarette tobacco products on the survival of patients with p16-positive oropharyngeal cancers is undefined. While there are reportedly increased risks of head and neck cancer associated with sustained heavy cigar and pipe use (Wyss 2013), such sustained use of non-cigarette products is unusual and does not appear to convey added risk with synchronous cigarette smoking. Cigar and pipe tobacco consumption is therefore not included in calculating the lifetime pack-years. Marijuana consumption is likewise not considered in this calculation. There is no clear scientific evidence regarding the role of chewing tobacco-containing products in this disease, although this is possibly more concerning given the proximity of the oral cavity and oropharynx. In any case, investigators are discouraged from enrolling patients with a history of very sustained use (such as several years or more) of non-cigarette tobacco products alone
* Zubrod performance status of 0-1 within 14 days prior to registration
* Age >= 18
* Absolute neutrophil count >= 1,500/mcL (within 14 days prior to registration)
* Platelets >= 100,000/mcL (within 14 days prior to registration)
* Hemoglobin >= 8.0 g/dL (within 14 days prior to registration) (Note: use of transfusion or other intervention to achieve hemoglobin [Hgb] >= 8.0 g/dL is acceptable)
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (within 14 days prior to registration)
* Aspartate aminotransferase (AST)(serum glutamic-oxaloacetic transaminase [SGOT]) or alanine aminotransferase (ALT)(serum glutamate pyruvate transaminase [SGPT]) =< 3.0 x institutional ULN (within 14 days prior to registration)
* Serum creatinine =< 1.5 x ULN OR creatinine clearance (CrCl) >= 50 mL/min (if using the Cockcroft-Gault formula) (within 14 days prior to registration)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated

  * Note: Known positive test for hepatitis B virus surface antigen (HBV sAg) indicating acute or chronic infection would make the patient ineligible unless the viral load becomes undetectable on suppressive therapy. Patients who are immune to hepatitis B (anti-hepatitis B surface antibody positive) are eligible (e.g. patients immunized against hepatitis B)
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment for the hepatitis, they are eligible if they have an undetectable HCV viral load.

  * Note: Known positive test for hepatitis C virus ribonucleic acid (HCV RNA) indicating acute or chronic infection would make the patient ineligible unless the viral load becomes undetectable on suppressive therapy
* For women of childbearing potential (WOCBP), negative serum or urine pregnancy test within 24 hours prior to registration

  * Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal. Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes. In addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL
* Women of childbearing potential (WOCBP) and men who are sexually active with WOCBP must be willing to use an adequate method of contraception during and after treatment
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry
* Only English, Spanish, or French speaking patients are eligible to participate as these are the only languages for which the mandatory dysphagia-related patient reported instrument (MDADI) is available

Exclusion Criteria:

* Clinical stages T0; T4; T1-2, N0; or any N2 (AJCC, 8th ed)
* Recurrent disease
* Definitive clinical or radiologic evidence of metastatic disease or adenopathy below the clavicles
* Cancers considered to be from an oral cavity site (oral tongue, floor mouth, alveolar ridge, buccal or lip), or the nasopharynx, hypopharynx, or larynx, even if p16-positive, or histologies of adenosquamous, verrucous, or spindle cell carcinomas
* Carcinoma of the neck of unknown primary site origin (T0 is ineligible, even if p16-positive)
* Radiographically matted nodes, defined as 3 abutting nodes with loss of the intervening fat plane
* Supraclavicular nodes, defined as nodes centered below the level of the cricoid cartilage
* Gross total excision of both primary and nodal disease; this includes tonsillectomy, local excision of primary site, and nodal excision that removes all clinically and radiographically evident disease. In other words, to participate in this protocol, the patient must have clinically or radiographically evident gross disease for which disease response can be assessed
* Patients with simultaneous primary cancers or separate bilateral primary tumor sites are excluded with the exception of patients with bilateral tonsil cancers
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 1095 days (3 years) (of note, the exclusion applies only for invasive cancers such that carcinoma in situ of the breast, oral cavity, or cervix are all permissible)
* Prior systemic chemotherapy for the study cancer; note that prior chemotherapy for a different cancer is allowable
* Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Severe, active co-morbidity defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days of registration
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition with immune compromise greater than that noted; note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because the treatments involved in this protocol may be significantly immunosuppressive. Protocol-specific requirements may also exclude immuno-compromised patients
  * Condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of registration. Inhaled or topical steroids and adrenal replacement doses < 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease
  * Patients with active autoimmune disease requiring systemic treatment (i.e. disease modifying agents, corticosteroids, or immunosuppressive drugs) should be excluded. These include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), rheumatoid arthritis, connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease
  * Note: Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Patients who are pregnant, nursing, or expecting to conceive or father children
* Prior allergic reaction to cisplatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2025-12-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sue S Yom, Principal Investigator — NRG Oncology
Locations (494):
- United States (493):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - Kaiser Permanente-Deer Valley Medical Center, Antioch, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Kaiser Permanente Dublin, Dublin, California
  - UC San Diego Health System - Encinitas, Encinitas, California
  - Kaiser Permanente-Fremont, Fremont, California
  - Fresno Cancer Center, Fresno, California
  - Kaiser Permanente-Fresno, Fresno, California
  - City of Hope at Irvine Lennar, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - City of Hope Antelope Valley, Lancaster, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Kaiser Permanente-Modesto, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Kaiser Permanente Oakland-Broadway, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente-Rancho Cordova Cancer Center, Rancho Cordova, California
  - Kaiser Permanente- Marshall Medical Offices, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Rohnert Park Cancer Center, Rohnert Park, California
  - Kaiser Permanente-Roseville, Roseville, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - The Permanente Medical Group-Roseville Radiation Oncology, Roseville, California
  - Kaiser Permanente Downtown Commons, Sacramento, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - South Sacramento Cancer Center, Sacramento, California
  - UC San Diego Medical Center - Hillcrest, San Diego, California
  - Naval Medical Center -San Diego, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - UCSF Medical Center-Mission Bay, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Stanford Cancer Center South Bay, San Jose, California
  - Kaiser Permanente San Leandro, San Leandro, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Kaiser San Rafael-Gallinas, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - City of Hope South Pasadena, South Pasadena, California
  - Kaiser Permanente Cancer Treatment Center, South San Francisco, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - City of Hope South Bay, Torrance, California
  - Torrance Memorial Physician Network - Cancer Care, Torrance, California
  - Torrance Memorial Medical Center, Torrance, California
  - City of Hope Upland, Upland, California
  - Kaiser Permanente Medical Center-Vacaville, Vacaville, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - Rocky Mountain Regional VA Medical Center, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers-Boulder, Boulder, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - UCHealth Memorial Hospital Central, Colorado Springs, Colorado
  - Memorial Hospital North, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Cancer Care and Hematology-Fort Collins, Fort Collins, Colorado
  - UCHealth Greeley Hospital, Greeley, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Medical Center of the Rockies, Loveland, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Hartford Hospital, Hartford, Connecticut
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Springs, Coral Springs, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center - McKinley Campus, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Moffitt Cancer Center at Wesley Chapel, Wesley Chapel, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Hawaii Cancer Care Inc - Waterfront Plaza, Honolulu, Hawaii
  - Queen's Cancer Cenrer - POB I, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - Queen's Cancer Center - Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kaiser Permanente Moanalua Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Cancer Care - Westridge, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Rush-Copley Medical Center, Aurora, Illinois
  - Advocate Good Shepherd Hospital, Barrington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - AMG Crystal Lake - Oncology, Crystal Lake, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Advocate Good Samaritan Hospital, Downers Grove, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Illinois CancerCare - Washington, Washington, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Broadlawns Medical Center, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Methodist West Hospital, West Des Moines, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - The University of Kansas Cancer Center - Olathe, Olathe, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - University of Kansas Health System Saint Francis Campus, Topeka, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Norton Hospital Pavilion and Medical Campus, Louisville, Kentucky
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Norton Brownsboro Hospital and Medical Campus, Louisville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Louisiana Hematology Oncology Associates LLC, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - MaineHealth Coastal Cancer Treatment Center, Bath, Maine
  - MaineHealth Maine Medical Center - Biddeford, Biddeford, Maine
  - MaineHealth Maine Medical Center - Portland, Portland, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - MaineHealth Cancer Care and IV Therapy - Sanford, Sanford, Maine
  - MaineHealth Cancer Care Center of York County, Sanford, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - MaineHealth Cancer Care and IV Therapy - South Portland, South Portland, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - UM Upper Chesapeake Medical Center, Bel Air, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Trinity Health Saint Joseph Mercy Hospital Ann Arbor, Ann Arbor, Michigan
  - McLaren Cancer Institute-Bay City, Bay City, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health Medical Center - Brighton, Brighton, Michigan
  - Henry Ford Cancer Institute-Downriver, Brownstown, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health Medical Center - Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - Chelsea Hospital, Chelsea, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - McLaren Cancer Institute-Clarkston, Clarkston, Michigan
  - Henry Ford Macomb Hospital-Clinton Township, Clinton Township, Michigan
  - Henry Ford Medical Center-Fairlane, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - McLaren Cancer Institute-Flint, Flint, Michigan
  - Singh and Arora Hematology Oncology PC, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Corewell Health Grand Rapids Hospitals - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Karmanos Cancer Institute at McLaren Greater Lansing, Lansing, Michigan
  - Mid-Michigan Physicians-Lansing, Lansing, Michigan
  - University of Michigan Health - Sparrow Lansing, Lansing, Michigan
  - McLaren Cancer Institute-Lapeer Region, Lapeer, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - McLaren Cancer Institute-Macomb, Mount Clemens, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Henry Ford Medical Center-Columbus, Novi, Michigan
  - McLaren Cancer Institute-Northern Michigan, Petoskey, Michigan
  - McLaren-Port Huron, Port Huron, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - Henry Ford Macomb Health Center - Shelby Township, Shelby, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Sanford Joe Lueken Cancer Center, Bemidji, Minnesota
  - Essentia Health Saint Joseph's Medical Center, Brainerd, Minnesota
  - Essentia Health - Deer River Clinic, Deer River, Minnesota
  - Essentia Health Cancer Center, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Essentia Health Hibbing Clinic, Hibbing, Minnesota
  - Coborn Cancer Center at Saint Cloud Hospital, Saint Cloud, Minnesota
  - Essentia Health Sandstone, Sandstone, Minnesota
  - Essentia Health Virginia Clinic, Virginia, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Parkland Health Center - Farmington, Farmington, Missouri
  - Freeman Health System, Joplin, Missouri
  - University of Kansas Cancer Center - North, Kansas City, Missouri
  - University of Kansas Cancer Center - Lee's Summit, Lee's Summit, Missouri
  - University of Kansas Cancer Center at North Kansas City Hospital, North Kansas City, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - CHI Health Good Samaritan, Kearney, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Sands Cancer Center, Canandaigua, New York
  - Noyes Memorial Hospital/Myers Cancer Center, Dansville, New York
  - Upstate Cancer Center at Oswego, Oswego, New York
  - Highland Hospital, Rochester, New York
  - University of Rochester, Rochester, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - SUNY Upstate Medical Center-Community Campus, Syracuse, New York
  - Upstate Cancer Center at Verona, Verona, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Atrium Health Pineville/LCI-Pineville, Charlotte, North Carolina
  - Atrium Health University City/LCI-University, Charlotte, North Carolina
  - Levine Cancer Institute-Ballantyne, Charlotte, North Carolina
  - Wake Forest University at Clemmons, Clemmons, North Carolina
  - Atrium Health Cabarrus/LCI-Concord, Concord, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Novant Health Cancer Institute - Huntersville, Huntersville, North Carolina
  - Novant Health Presbyterian Medical Center Huntersville, Huntersville, North Carolina
  - Novant Health Cancer Institute - Kernersville, Kernersville, North Carolina
  - Novant Health Cancer Institute - Matthews, Matthews, North Carolina
  - Atrium Health Union/LCI-Union, Monroe, North Carolina
  - Novant Health Cancer Institute - Mooresville, Mooresville, North Carolina
  - Novant Health Cancer Institute - Mount Airy, Mount Airy, North Carolina
  - Novant Health Cancer Institute - Wilkesboro, North Wilkesboro, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hospital, Pinehurst, North Carolina
  - Novant Health Cancer Institute - Rowan, Salisbury, North Carolina
  - Novant Health Cancer Institute - Statesville, Statesville, North Carolina
  - Wake Forest Baptist Health - Hematology Oncology - Statesville, Statesville, North Carolina
  - Novant Cancer Institute Radiation Oncology - Supply, Supply, North Carolina
  - Novant Health Cancer Institute - Thomasville, Thomasville, North Carolina
  - Wake Forest Baptist Health - Wilkes Medical Center, Wilkesboro, North Carolina
  - Novant Health Cancer Institute Radiation Oncology - Wilmington, Wilmington, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Novant Health Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Summa Health System - Akron Campus, Akron, Ohio
  - UH Seidman Cancer Center at UH Avon Health Center, Avon, Ohio
  - Summa Health System - Barberton Campus, Barberton, Ohio
  - Geauga Hospital, Chardon, Ohio
  - University of Cincinnati Cancer Center-UC Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Cleveland Clinic Cancer Center Mansfield, Mansfield, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Summa Health Medina Medical Center, Medina, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - UH Seidman Cancer Center at Southwest General Hospital, Middleburg Heights, Ohio
  - University Hospitals Parma Medical Center, Parma, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - University Hospitals Portage Medical Center, Ravenna, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Cleveland Clinic Cancer Center Strongsville, Strongsville, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Mercy Health Sylvania Radiation Oncology Center, Toledo, Ohio
  - University of Cincinnati Cancer Center-West Chester, West Chester, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - UHHS-Westlake Medical Center, Westlake, Ohio
  - Cleveland Clinic Wooster Family Health and Surgery Center, Wooster, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Clackamas Radiation Oncology Center, Clackamas, Oregon
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Providence Willamette Falls Medical Center, Oregon City, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC Altoona, Altoona, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Carlisle Regional Cancer Center, Carlisle, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Fox Chase Cancer Center - East Norriton Hospital Outpatient Center, East Norriton, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - UPMC Hillman Cancer Center Erie, Erie, Pennsylvania
  - UPMC Cancer Center at UPMC Horizon, Farrell, Pennsylvania
  - Fox Chase Cancer Center Buckingham, Furlong, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - UPMC Pinnacle Cancer Center/Community Osteopathic Campus, Harrisburg, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC Hillman Cancer Center at Rocco And Nancy Ortenzio Cancer Pavilion, Mechanicsburg, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - UPMC Cancer Center - Monroeville, Monroeville, Pennsylvania
  - UPMC Hillman Cancer Center in Coraopolis, Moon Township, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Geisinger Cancer Services-Pottsville, Pottsville, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Divine Providence Hospital, Williamsport, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - UPMC Memorial, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Gibbs Cancer Center-Gaffney, Gaffney, South Carolina
  - Tidelands Georgetown Memorial Hospital, Georgetown, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Gibbs Cancer Center-Pelham, Greer, South Carolina
  - Rock Hill Radiation Therapy Center, Rock Hill, South Carolina
  - Levine Cancer Institute-Rock Hill, Rock Hill, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Spartanburg Medical Center, Spartanburg, South Carolina
  - SMC Center for Hematology Oncology Union, Union, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - The West Clinic - Wolf River, Germantown, Tennessee
  - University of Tennessee - Knoxville, Knoxville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - The Don and Sybil Harrington Cancer Center, Amarillo, Texas
  - American Fork Hospital / Huntsman Intermountain Cancer Center, American Fork, Utah
  - Farmington Health Center, Farmington, Utah
  - Logan Regional Hospital, Logan, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Riverton Hospital, Riverton, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Saint George Regional Medical Center, St. George, Utah
  - Dartmouth Cancer Center - North, Saint Johnsbury, Vermont
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Inova Fair Oaks Hospital, Fairfax, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Valley Medical Center, Renton, Washington
  - Swedish Medical Center-Ballard Campus, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Providence Saint Mary Regional Cancer Center, Walla Walla, Washington
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Ascension Saint Elizabeth Hospital, Appleton, Wisconsin
  - Duluth Clinic Ashland, Ashland, Wisconsin
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Elmbrook Campus, Brookfield, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Ascension Calumet Hospital, Chilton, Wisconsin
  - HSHS Sacred Heart Hospital, Eau Claire, Wisconsin
  - Ascension Saint Francis - Reiman Cancer Center, Franklin, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Franklin, Franklin, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Essentia Health-Hayward Clinic, Hayward, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Johnson Creek, Johnson Creek, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Froedtert Menomonee Falls Hospital, Menomonee Falls, Wisconsin
  - Ascension Columbia Saint Mary's Hospital Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Ascension Southeast Wisconsin Hospital - Saint Joseph Campus, Milwaukee, Wisconsin
  - Ascension Columbia Saint Mary's Hospital - Milwaukee, Milwaukee, Wisconsin
  - Ascension Saint Francis Hospital, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Ascension Mercy Hospital, Oshkosh, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Ascension All Saints Hospital, Racine, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Aspirus Cancer Care - James Beck Cancer Center, Rhinelander, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Essentia Health-Spooner Clinic, Spooner, Wisconsin
  - Aspirus Cancer Care - Stevens Point, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Essentia Health Saint Mary's Hospital - Superior, Superior, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Ascension Medical Group Southeast Wisconsin - Mayfair Road, Wauwatosa, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Froedtert West Bend Hospital/Kraemer Cancer Center, West Bend, Wisconsin
  - Aspirus Cancer Care - Wisconsin Rapids, Wisconsin Rapids, Wisconsin
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm II (Reduced RT+ Cisplatin): Patients undergo reduced dose RT as 60 Gy IMRT or IGRT QD over 5 fractions per week and receive 100 mg/m^2/day cisplatin IV over 30-60 minutes on days 1 and 22. Treatment continues for 6 weeks in the absence of disease progression or unacceptable toxicity. Patients receive FDG and undergo PET/CT or CT during screening and during follow up, and undergo MRI during follow up. Patients may also undergo tissue biopsy and blood sample collection throughout the study.
Period: Overall Study
Arm/Group | Arm I (Standard RT + Cisplatin) | Arm II (Reduced RT+ Cisplatin) | Arm III (Reduced RT + Nivolumab)
Started (Randomized) | 136 | 116 | 132
Adverse Event Populaton (Started protocol treatment.) | 123 | 112 | 123
Completed (Participants contributing data to any results are considered to have completed the study.) | 136 | 116 | 132
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Standard RT + Cisplatin) | Arm II (Reduced RT+ Cisplatin) | Arm III (Reduced RT + Nivolumab) | Total
Number analyzed (Participants) | 136 | 116 | 132 | 384
Age, Continuous [Median (Full Range); unit: years] | 60 [37 to 81] | 61 [41 to 79] | 60.5 [36 to 78] | 60 [36 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 13 | 36
  Male | 124 | 105 | 119 | 348
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 9 | 7 | 20
  Not Hispanic or Latino | 124 | 104 | 120 | 348
  Unknown or Not Reported | 8 | 3 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Asian | 3 | 3 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 6 | 6 | 16
  White | 118 | 102 | 116 | 336
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 10 | 4 | 5 | 19
Zubrod performance status [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound; 5 = Death
  Participants
    0 | 118 | 102 | 117 | 337
    1 | 18 | 14 | 15 | 47
Smoking history [Count of Participants; unit: Participants]
  Never | 108 | 93 | 104 | 305
  Former | 28 | 22 | 28 | 78
  Current | 0 | 1 | 0 | 1
Pack-years [Count of Participants; unit: Participants] — A way to measure the amount a person has smoked over a long period of time. It is calculated by multiplying the number of packs of cigarettes smoked per day by the number of years the person has smoked. Note, only the person's age when smoking started and stopped was collected, therefore if a person started and stopped at the same age, then pack-years would be computed as zero even though the person had smoked during that year.
  Participants
    0 | 109 | 93 | 104 | 306
    >0 to ≤10 | 27 | 23 | 28 | 78
Primary tumor site [Count of Participants; unit: Participants]
  Oropharynx NOS | 16 | 12 | 10 | 38
  Tonsillar fossa, tonsil | 68 | 55 | 65 | 188
  Base of tongue | 51 | 46 | 54 | 151
  Pharyngeal oropharynx | 1 | 3 | 3 | 7
p16-positive status [Count of Participants; unit: Participants] — The biomarker p16 is used as a surrogate marker for human papillomavirus (HPV) infections and is a known prognostic factor in some head and neck cancers.
  Participants | 136 | 116 | 132 | 384
T stage, clinical (AJCC 8) [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 8th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b.
  Participants
    T0 | 1 | 0 | 0 | 1
    T1 | 50 | 39 | 51 | 140
    T2 | 68 | 57 | 61 | 186
    T3 | 17 | 20 | 20 | 57
N stage, clinical (AJCC 8) [Count of Participants; unit: Participants] — Regional lymph nodes staging per American Joint Committee on Cancer (AJCC) 8th ed. refers to the number and/or extent of spread of lymph nodes that contain cancer. N0 means lymph nodes aren't involved. A higher number means the cancer is in more lymph nodes, farther away from the original tumor. NX means the lymph nodes cannot be assessed.
  Participants
    N0 | 5 | 4 | 4 | 13
    N1 | 131 | 112 | 126 | 369
    N2 | 0 | 0 | 1 | 1
    N3 | 0 | 0 | 1 | 1
M stage M0, clinical (AJCC 8) [Count of Participants; unit: Participants] — Metastasis stage per the American Joint Committee on Cancer (AJCC) 8th ed. refers to the spread of the cancer to organs and tissues in other parts of the body. M0 = No distant metastasis; M1 = Distant metastasis; MX = Distant metastasis cannot be assessed.
  Participants | 136 | 116 | 132 | 384
Stage group, clinical (AJCC 8) [Count of Participants; unit: Participants] — Overall cancer stage per American Joint Committee on Cancer (AJCC) 8th ed. combines tumor (T), regional lymph node (N), and distant metastasis (M) staging to determine an overall stage of 0, I, II, III, or IV, ranging from least to most advanced, respectively. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. The higher the number after the N, the greater the involvement of regional lymph nodes. M0 indicates no distant metastasis.
  Participants
    I (T0-2,N0-1,M0) | 119 | 96 | 111 | 326
    II (T0-2,N2,M0 or T3,N0-2,M0) | 17 | 20 | 20 | 57
    III (T0-3, N3, M0) | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) (Phase II) (Percentage of Participants Alive Without Progression)
Description: Progression is defined as local-regional progression or recurrence, distant metastasis, death due to any reason, salvage surgery of primary with tumor present/unknown, salvage neck dissection with tumor present/unknown, > 20 weeks from end of radiation therapy. Progression-free survival rates are estimated using the Kaplan-Meier method, censoring participants alive at time of analysis.
  The primary phase IIR endpoint is tested using a confidence interval (CI) approach with each experimental arm compared to the standard arm (Arm 1).
Time Frame: From randomization to first progression or last follow-up. Maximum follow-up at the time of analysis was 4.6 years. The 1- and 2-year estimates are reported.
Population: Randomized phase II participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Standard RT + Cisplatin) | Arm II (Reduced RT+ Cisplatin) | Arm III (Reduced RT + Nivolumab)
Number analyzed (Participants) | 136 | 116 | 132
percentage of participants
  1 year | 99.1 [97.3 to 100] | 96.4 [93.0 to 99.9] | 96.6 [93.4 to 99.9]
  2 years | 98.1 [95.4 to 100] | 88.6 [82.4 to 94.7] | 90.3 [84.5 to 96.1]
Statistical Analysis 1: Comparison: Arm I (Standard RT + Cisplatin) vs Arm II (Reduced RT+ Cisplatin); The null hypothesis (H0) for each comparison in phase II will be rejected if the 90% upper confidence of the hazard ratio (HR) (experimental arm / standard arm) is less than HR=2.4; Test type: Non-Inferiority — Estimated 9-month PFS = 96.5% and lower acceptable threshold = 91.8%, resulting in a non-inferiority margin of 4.7%. H0: HR = 2.4; alternative hypothesis (HA): HR=1.0. One-sided type I error rate of 10% (20% after Bonferroni adjustment for each experimental arm comparison), 80% power, 24 months of accrual with 1 year of additional follow-up, and 1% increasing yearly rate of drop-out up to 3%, a log rank test requires 22 events from 266 patients per comparison resulting in 133 patients per arm; Hazard Ratio (HR) = 7.42, 90% CI 1-sided [upper limit 19.46] — Reference level = Arm 1
Statistical Analysis 2: Comparison: Arm I (Standard RT + Cisplatin) vs Arm III (Reduced RT + Nivolumab); [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 5.55, 90% CI 1-sided [upper limit 14.85] — Reference level = Arm 1

2. Primary Outcome: Progression-free Survival (Phase III) (Percentage of Participants Alive Without Progression)
Description: Progression is defined as local-regional progression or recurrence, distant metastasis, death due to any reason, salvage surgery of primary with tumor present/unknown, salvage neck dissection with tumor present/unknown, > 20 weeks from end of radiation therapy. Progression-free survival rates are estimated using the Kaplan-Meier method, censoring participants alive at time of analysis.
Time Frame: From randomization to first progression or last follow-up. Maximum follow-up was 4.6 years.
Population: Randomized phase III participants. (Phase III component did not and will not open.)
Arm/Group | Arm I (Standard RT + Cisplatin) | Arm II (Reduced RT+ Cisplatin) | Arm III (Reduced RT + Nivolumab)
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: MD Anderson Dysphagia Inventory (MDADI) Global Quality of Life (QOL) Score
Description: The M. D. Anderson Dysphagia Inventory (MDADI) assesses how patients view their swallowing ability as a result of treatment and how this affects their QOL. It consists of a global quality of life question and a functional, emotional, and physical subscale. The global QOL question ranges from 1 to 5 and multiplied by 20 to obtain a score with a range of 0 to 100. Higher scores indicate better functioning.
Time Frame: Baseline to two years
Population: Randomized phase III participants. (Phase III component did not and will not open.)
Arm/Group | Arm I (Standard RT + Cisplatin) | Arm II (Reduced RT+ Cisplatin) | Arm III (Reduced RT + Nivolumab)
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Locoregional Failure (Percentage of Participants With Locoregional Failure)
Description: Locoregional failure is defined as local-regional progression or recurrence, death due to study cancer or unknown causes, salvage neck dissection with tumor present/unknown. Locoregional failure rates are estimated the cumulative incidence method, treating distant metastasis and death due to any reason other than study cancer or unknown as competing risks, and otherwise censoring participants alive at time of analysis. Each experimental arm is compared to the standard arm (Arm I).
Time Frame: From randomization to first failure, competing event, or last known follow-up, whichever occurs first. Maximum follow-up at the time of analysis was 4.6 years. The 1- and 2-year estimates are reported.
Population: Randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Standard RT + Cisplatin) | Arm II (Reduced RT+ Cisplatin) | Arm III (Reduced RT + Nivolumab)
Number analyzed (Participants) | 136 | 116 | 132
percentage of participants
  1 year | 0.0 [NA to NA] — Cannot be calculated for zero. | 2.7 [0.7 to 7.0] | 1.7 [0.3 to 5.4]
  2 years | 0.0 [NA to NA] — Cannot be calculated for zero. | 6.5 [2.8 to 12.2] | 5.0 [1.8 to 10.6]
Statistical Analysis 1: Comparison: Arm I (Standard RT + Cisplatin) vs Arm II (Reduced RT+ Cisplatin); Test type: Superiority; Hazard Ratio (HR) = 20.56, 95% CI 2-sided [1.05 to 403.31] — Cause-specific; reference level = Arm 1
Statistical Analysis 2: Comparison: Arm I (Standard RT + Cisplatin) vs Arm III (Reduced RT + Nivolumab); Test type: Superiority; Hazard Ratio (HR) = 12.87, 95% CI 2-sided [0.58 to 287.93] — Reference level = Arm 1

5. Secondary Outcome: Distant Failure (Percentage of Participants With Distant Failure)
Description: Distant failure is defined as the occurrence of distant metastasis. Distant failure rates are estimated the cumulative incidence method, treating local-regional progression or recurrence, death due to any reason, salvage neck dissection with tumor present/unknown as competing risks, and otherwise censoring participants alive at time of analysis. Each experimental arm is compared to the standard arm (Arm I).
Time Frame: as for outcome 4
Population: Randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Standard RT + Cisplatin) | Arm II (Reduced RT+ Cisplatin) | Arm III (Reduced RT + Nivolumab)
Number analyzed (Participants) | 136 | 116 | 132
percentage of participants
  Year 1 | 0.9 [0.1 to 4.5] | 0.0 [NA to NA] — Cannot be calculated for zero. | 0.8 [0.1 to 4.2]
  Year 2 | 1.9 [0.4 to 6.2] | 4.1 [1.3 to 9.4] | 2.9 [0.8 to 7.8]
Statistical Analysis 1: Comparison: Arm I (Standard RT + Cisplatin) vs Arm II (Reduced RT+ Cisplatin); Test type: Superiority; Cox Proportional Hazard = 1.78, 95% CI 2-sided [0.34 to 9.46] — Cause-specific; reference level = Arm 1
Statistical Analysis 2: Comparison: Arm I (Standard RT + Cisplatin) vs Arm III (Reduced RT + Nivolumab); Test type: Superiority; Cox Proportional Hazard = 1.43, 95% CI 2-sided [0.24 to 8.45] — Cause-specific; reference level = Arm 1

6. Secondary Outcome: Overall Survival (Percentage of Participants Alive)
Description: Survival rates are estimated using the Kaplan-Meier method, censoring participants alive at time of analysis.
Time Frame: From randomization to death from any cause or last follow-up. Maximum follow-up at the time of analysis was 4.6 years. The 1- and 2-year estimates are reported.
Population: Randomized participants
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Arm I (Standard RT + Cisplatin) | Arm II (Reduced RT+ Cisplatin) | Arm III (Reduced RT + Nivolumab)
Number analyzed (Participants) | 136 | 116 | 132
Percent of participants
  1 year | 100 [NA to NA] — Cannot be calculated for 100. | 99.1 [97.4 to 100] | 99.2 [97.5 to 100]
  2 year | 99.0 [97.0 to 100] | 98.0 [95.2 to 100] | 96.1 [92.3 to 99.9]
Statistical Analysis 1: Comparison: Arm I (Standard RT + Cisplatin) vs Arm II (Reduced RT+ Cisplatin); Test type: Superiority; Hazard Ratio (HR) = 5.58, 95% CI 2-sided [0.67 to 46.41] — Reference level = Arm 1
Statistical Analysis 2: Comparison: Arm I (Standard RT + Cisplatin) vs Arm III (Reduced RT + Nivolumab); Test type: Superiority; Hazard Ratio (HR) = 4.87, 95% CI 2-sided [0.57 to 41.74] — Reference level = Arm 1

7. Secondary Outcome: Number of Participants by Highest Grade Adverse Event Reported
Description: Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grades adverse event severity as follows: 1 = mild, 2 = moderate, 3 = severe, 4 = life-threatening, 5 = death related to adverse event. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data.
Time Frame: From randomization to last known follow-up. Maximum follow-up at the time of analysis was 4.6 years.
Population: Randomized and started protocol treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Standard RT + Cisplatin) | Arm II (Reduced RT+ Cisplatin) | Arm III (Reduced RT + Nivolumab)
Number analyzed (Participants) | 123 | 112 | 123
Participants
  Grade 1 | 3 | 4 | 4
  Grade 2 | 37 | 27 | 38
  Grade 3 | 68 | 66 | 72
  Grade 4 | 15 | 15 | 8

8. Secondary Outcome: Hearing
Description: Measured as Hearing Handicap Inventory for Adults-Screening (HHIA-S).
Time Frame: Baseline up to 24 months from end of radiation therapy (RT)
Reporting Status: Not Posted, anticipated posting 2027-02

9. Secondary Outcome: Quality of Life
Description: Measured by the European Organization for Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire (QLQ)30.
Time Frame: Baseline up to 24 months from end of RT
Reporting Status: Not Posted, anticipated posting 2027-02

10. Secondary Outcome: Fludeoxyglucose F-18 (FDG)-Positron Emission Tomography (PET)/Computed Tomography (CT) Locoregional Control
Description: Will be associated with PFS.
Time Frame: Up to 6 years
Reporting Status: Not Posted, anticipated posting 2027-02

11. Secondary Outcome: Negative Predictive Value of Post-RT FDG-PET/CT for Locoregional Control
Description: The negative predictive value of FDG-PET/CT for locoregional control will be estimated using binomial proportions and confidence intervals based on normal approximation.
Time Frame: At 1 and 2 years
Reporting Status: Not Posted, anticipated posting 2027-02

12. Secondary Outcome: Negative Predictive Value of Post-RT FDG-PET/CT for PFS
Description: The negative predictive value of FDG-PET/CT PFS will be estimated using binomial proportions and confidence intervals based on normal approximation.
Time Frame: At 1 and 2 years
Reporting Status: Not Posted, anticipated posting 2027-02

13. Secondary Outcome: Incidence of Adverse Events
Description: Measured using Patient-Reported Outcomes (PRO)-CTCAE. For each symptom, counts and frequencies will be provided for the worst score experienced by the patient by treatment arm. The proportion of patients with scores >= 1 and >= 3 will be compared between groups using a Chi-square test, or Fisher's exact test if cell frequencies are < 5, using a significance level of 0.05. Analysis of changes in patient reported outcomes over time will analyzed by fitting generalized estimating equations (GEE) models using a logit link (dichotomizing the symptom scores as 0 vs. > 1 and 0-2 vs. 3-4) with time of assessment, treatment arm, and treatment-by-time interaction terms in the model.
Time Frame: Up to 6 years
Reporting Status: Not Posted, anticipated posting 2027-02

14. Other Pre Specified Outcome: Quality of Life
Description: Measured by EuroQol-5 Dimensional- 5 Level (EQ-5D-5L).
Time Frame: Baseline up to 24 months from end of RT
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Swallowing Physiology
Description: Measured by a Modified Barium Swallow (MBS) test. The proportion of aspiration for each arm will be estimated assuming a binomial distribution and between arm comparison will be performed using a Fisher's exact test.
Time Frame: Up to 6 years
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Locoregional Control for Patients With Post-RT FDG-PET/CT
Description: Locoregional control rates will be compared between negative and positive/undetermined patients. Cox proportional hazards models will be used to determine whether there are differences between these two groups, while adjusting for treatment arm and other covariates (cause-specific Cox models for locoregional failure).
Time Frame: At 12-14 weeks post-RT
Reporting Status: Not Posted

17. Other Pre Specified Outcome: PFS for Patients With Post-RT FDG-PET/CT
Description: PFS rates will be compared between negative and positive/undetermined patients. Cox proportional hazards models will be used to determine whether there are differences between these two groups, while adjusting for treatment arm and other covariates (cause-specific Cox models for locoregional failure).
Time Frame: At 12-14 weeks post-RT
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From randomization to death or last follow-up. Maximum follow-up at the time of analysis was 4.6 years.
Description: All-cause mortality was assessed in randomized participants. Adverse events were assessed in randomized participants who started protocol treatment.
Arm/Group | Arm I (Standard RT + Cisplatin) | Arm II (Reduced RT+ Cisplatin) | Arm III (Reduced RT + Nivolumab)
All-Cause Mortality (participants affected / at risk) | 1/136 | 6/116 | 5/132
Serious Adverse Events (participants affected / at risk) | 49/123 | 32/112 | 34/123
Other Adverse Events (participants affected / at risk) | 123/123 | 111/112 | 122/123
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Standard RT + Cisplatin) (N=123) | Arm II (Reduced RT+ Cisplatin) (N=112) | Arm III (Reduced RT + Nivolumab) (N=123)
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 2 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 2
Testosterone deficiency (Endocrine disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 2
Colitis (Gastrointestinal disorders) | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 5 | 5 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 5 | 6 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 12 | 4 | 1
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 13 | 9 | 7
Nausea (Gastrointestinal disorders) | 13 | 14 | 5
Obstruction gastric (Gastrointestinal disorders) | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 1 | 3 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 5 | 4
Edema limbs (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 2 | 3 | 0
Fever (General disorders) | 2 | 0 | 1
General disorders and administration site conditions - Other (General disorders) | 1 | 0 | 1
Localized edema (General disorders) | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0
Neck edema (General disorders) | 0 | 0 | 1
Pain (General disorders) | 2 | 0 | 0
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 0 | 1 | 0
Immune system disorders - Other (Immune system disorders) | 0 | 0 | 2
Infections and infestations - Other (Infections and infestations) | 1 | 1 | 2
Lung infection (Infections and infestations) | 0 | 0 | 3
Mucosal infection (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 2
Thrush (Infections and infestations) | 5 | 4 | 4
Tooth infection (Infections and infestations) | 0 | 0 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 6 | 5 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Injury, poisoning and procedural complications - Other (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 0 | 0 | 1
CPK increased (Investigations) | 0 | 0 | 1
Creatinine increased (Investigations) | 8 | 8 | 3
Neutrophil count decreased (Investigations) | 3 | 4 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Weight loss (Investigations) | 9 | 3 | 2
White blood cell decreased (Investigations) | 2 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 11 | 3 | 0
Dehydration (Metabolism and nutrition disorders) | 7 | 8 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 5 | 3 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 3 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 2
Dysphasia (Nervous system disorders) | 1 | 1 | 1
Headache (Nervous system disorders) | 2 | 0 | 2
Paresthesia (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 4 | 1
Chronic kidney disease (Renal and urinary disorders) | 0 | 2 | 0
Hematuria (Renal and urinary disorders) | 2 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 | 0 | 1
Hematoma (Vascular disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 3 | 0 | 1
Lymphedema (Vascular disorders) | 1 | 1 | 0
Thromboembolic event (Vascular disorders) | 4 | 2 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Standard RT + Cisplatin) (N=123) | Arm II (Reduced RT+ Cisplatin) (N=112) | Arm III (Reduced RT + Nivolumab) (N=123)
Anemia (Blood and lymphatic system disorders) | 52 | 53 | 33
Ear pain (Ear and labyrinth disorders) | 7 | 10 | 10
Hearing impaired (Ear and labyrinth disorders) | 33 | 34 | 10
Tinnitus (Ear and labyrinth disorders) | 75 | 66 | 28
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 15
Hypothyroidism (Endocrine disorders) | 5 | 2 | 25
Blurred vision (Eye disorders) | 7 | 4 | 5
Abdominal pain (Gastrointestinal disorders) | 13 | 7 | 10
Constipation (Gastrointestinal disorders) | 50 | 53 | 41
Diarrhea (Gastrointestinal disorders) | 16 | 16 | 19
Dry mouth (Gastrointestinal disorders) | 100 | 94 | 114
Dyspepsia (Gastrointestinal disorders) | 8 | 7 | 4
Dysphagia (Gastrointestinal disorders) | 87 | 68 | 86
Esophagitis (Gastrointestinal disorders) | 7 | 2 | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 9 | 9 | 8
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 5 | 12 | 4
Mucositis oral (Gastrointestinal disorders) | 92 | 78 | 92
Nausea (Gastrointestinal disorders) | 80 | 72 | 45
Oral pain (Gastrointestinal disorders) | 19 | 15 | 32
Salivary duct inflammation (Gastrointestinal disorders) | 9 | 6 | 5
Vomiting (Gastrointestinal disorders) | 37 | 32 | 19
Fatigue (General disorders) | 104 | 86 | 101
Neck edema (General disorders) | 4 | 4 | 10
Pain (General disorders) | 13 | 16 | 14
Thrush (Infections and infestations) | 15 | 16 | 19
Dermatitis radiation (Injury, poisoning and procedural complications) | 72 | 67 | 90
Alanine aminotransferase increased (Investigations) | 25 | 19 | 15
Alkaline phosphatase increased (Investigations) | 1 | 7 | 4
Aspartate aminotransferase increased (Investigations) | 9 | 10 | 17
Blood bilirubin increased (Investigations) | 6 | 6 | 7
Creatinine increased (Investigations) | 48 | 41 | 18
Investigations - Other (Investigations) | 4 | 8 | 6
Lymphocyte count decreased (Investigations) | 61 | 70 | 68
Neutrophil count decreased (Investigations) | 42 | 41 | 4
Platelet count decreased (Investigations) | 36 | 40 | 12
Thyroid stimulating hormone increased (Investigations) | 3 | 3 | 7
Weight loss (Investigations) | 78 | 84 | 91
White blood cell decreased (Investigations) | 55 | 51 | 24
Anorexia (Metabolism and nutrition disorders) | 45 | 44 | 48
Dehydration (Metabolism and nutrition disorders) | 17 | 16 | 12
Hypercalcemia (Metabolism and nutrition disorders) | 7 | 0 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 32 | 30 | 25
Hyperkalemia (Metabolism and nutrition disorders) | 6 | 6 | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 14 | 11 | 14
Hypocalcemia (Metabolism and nutrition disorders) | 8 | 15 | 5
Hypokalemia (Metabolism and nutrition disorders) | 24 | 16 | 14
Hypomagnesemia (Metabolism and nutrition disorders) | 18 | 17 | 4
Hyponatremia (Metabolism and nutrition disorders) | 37 | 33 | 25
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 9
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 8 | 5
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 3 | 4 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 13 | 12 | 15
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 8 | 2
Trismus (Musculoskeletal and connective tissue disorders) | 5 | 6 | 7
Dizziness (Nervous system disorders) | 19 | 11 | 13
Dysgeusia (Nervous system disorders) | 96 | 95 | 93
Headache (Nervous system disorders) | 14 | 22 | 23
Paresthesia (Nervous system disorders) | 6 | 6 | 5
Peripheral sensory neuropathy (Nervous system disorders) | 16 | 24 | 16
Anxiety (Psychiatric disorders) | 9 | 13 | 7
Depression (Psychiatric disorders) | 8 | 6 | 4
Insomnia (Psychiatric disorders) | 15 | 10 | 15
Chronic kidney disease (Renal and urinary disorders) | 8 | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 14 | 19
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 8 | 10
Hiccups (Respiratory, thoracic and mediastinal disorders) | 16 | 14 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 11 | 10 | 12
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 9
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 32 | 19 | 32
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 8
Sore throat (Respiratory, thoracic and mediastinal disorders) | 35 | 37 | 47
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 7 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 4 | 14
Rash acneiform (Skin and subcutaneous tissue disorders) | 4 | 2 | 7
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 5 | 10
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 6 | 4 | 7
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 1 | 7
Hypertension (Vascular disorders) | 20 | 22 | 17
Lymphedema (Vascular disorders) | 9 | 12 | 17

LIMITATIONS AND CAVEATS:
This phase II/III trial did not proceed to the phase III component, per the protocol. Arm 2 closed to accrual earlier than the other arms due to the timing of the futility analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT03952585/Prot_SAP_000.pdf
  • Informed Consent Form: Phase II Consent Document (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT03952585/ICF_001.pdf
  • Informed Consent Form: Phase III Consent Document (2023-08-21): https://cdn.clinicaltrials.gov/large-docs/85/NCT03952585/ICF_002.pdf